CLINICAL TRIAL: NCT06630546
Title: Trabecular Microbypass IStent in Patients with Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Ting Tsao (Other)
Responsible Party: Sponsor-Investigator, Yu-Ting Tsao, Clinical Doctor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202200593B0
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Primary Open Angle Glaucoma (POAG); Istent Inject W; Normal Tension Glaucoma (NTG)
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma | interventions — Mutagenesis, Insertional; Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- phacoemulsification combined with one trabecular micro-bypass stent implantation (phaco-iStent) (Experimental): In glaucoma patient who needed to receive cataract surgery, a standard phacoemulsification procedure was performed, along with the implantation of a foldable posterior chamber intraocular lens (PCIOL). Then, in this group, we further inserted a preloaded micro-bypass stent (model GTS100L) through the temporal corneal incision into the nasal Schlemm's canal and checked the position. Adequate intraocular pressure (IOP) was assessed by palpation at the end of the surgery.
  Interventions: Device: first generation iStent (Glaukos, San Clemente, CA, USA) insertion; Device: phacoemulsification
- phacoemulsification alone group (Active Comparator): In glaucoma patient who needed to receive cataract surgery, a standard phacoemulsification procedure was performed, along with the implantation of a foldable posterior chamber intraocular lens (PCIOL).
  Interventions: Device: phacoemulsification

INTERVENTIONS:
Device: first generation iStent (Glaukos, San Clemente, CA, USA) insertion — In glaucoma patient who needed to receive cataract surgery, a standard phacoemulsification procedure was performed, along with the implantation of a foldable posterior chamber intraocular lens (PCIOL). Then, in adequate patient who wish to receive iStent insertion, we further inserted a preloaded micro-bypass stent (model GTS100L) through the temporal corneal incision into the nasal Schlemm's canal and checked the position. Adequate intraocular pressure (IOP) was assessed by palpation at the end of the surgery.
  Arms: phacoemulsification combined with one trabecular micro-bypass stent implantation (phaco-iStent)
Device: phacoemulsification — A standard phacoemulsification procedure was performed, along with the implantation of a foldable posterior chamber intraocular lens (PCIOL).

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of phacoemulsification combined with one trabecular micro-bypass stent implantation (phaco-iStent) versus phacoemulsification alone in a Taiwanese population, as well as to investigate any differences in outcomes between patients with primary open angle glaucoma (POAG) and those with normal tension glaucoma (NTG). The main question it aims to answer is:

• How much do intraocular pressure (IOP) and the number of antiglaucoma medications change after iStent insertion, with subgroup analyses for POAG and NTG? Researchers will compare phacoemulsification combined with one trabecular micro-bypass stent implantation (phaco-iStent) versus phacoemulsification alone to see if IOP and the number of antiglaucoma medications decrease.

Participants will receive their regular phacoemulsification and decided whether to receive iStent by themselves.

ELIGIBILITY:
Inclusion Criteria:

Patients evaluated by a clinician who require cataract surgery or cataract surgery combined with iStent implantation due to concomitant glaucoma and cataracts.

Exclusion Criteria:

* Eyes that have previously undergone vitrectomy or retinal surgery.
* Patients with ocular surface inflammation (e.g., corneal ulcers, orbital cellulitis, etc.).
* Patients with hypotony (intraocular pressure <5 mmHg).
* Patients with a history of globe rupture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) in mmHg or percentage changes | From enrollment to the end of treatment at 18 months
  changes in IOP after the intervention
glaucoma medication changes in number | From enrollment to the end of treatment at 18 months
  glaucoma medication changes in number after the intervention
Visual acuity changes in LogMAR scale | From enrollment to the end of treatment at 18 months
  Visual acuity changes in LogMAR scale after the intervention in both group

SECONDARY OUTCOMES:
Complete success and qualified success | From enrollment to the end of treatment at 18 months
  Complete success was defined as postsurgical IOP of less than 21 mmHg without the use of any glaucoma medication, while qualified success was defined as postsurgical IOP not exceeding 21 mmHg with a reduction of one or more antiglaucoma agents compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital Linkou Branch, Taoyuan, No.5, Fuxing St., Guishan Dist.,, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Eligibility for Data Access:
  * Data will be shared with qualified researchers who provide a clear and scientifically valid research proposal.
  * Proposals that align with the objectives of the original study or are intended for research that could contribute to the scientific understanding of the field will be considered.
  Request Process:
  * Interested researchers can request data by sending an email that includes a description of the intended analyses and the purpose of the research.
  * No formal review process is required, but requests should demonstrate a valid scientific rationale for data access.
  Mechanism for Data Sharing:
  - Data will be shared via email. Once the request is received and approved, the data will be sent directly to the researcher.
  Time Frame for Data Access:
  - Data will be made available beginning 3 months and ending 3 years after the publication of results

REFERENCES:
- [Derived] Tsao YT, Yeh PH, Su WW. Comparison of Phacoemulsification Alone and With Trabecular Microbypass Stent in Primary Open-Angle Glaucoma and Normal-Tension Glaucoma: An 18-Month Outcome Study. J Ophthalmol. 2024 Nov 7;2024:4034215. doi: 10.1155/2024/4034215. eCollection 2024. PMID 39544960